CLINICAL TRIAL: NCT00328796
Title: Acupuncture or Local Anaesthetics for Pain Relief During Perineal Repair After Vaginal Delivery: A Randomised Controlled Trial
Brief Title: Acupuncture for Pain Relief During Perineal Repair After Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonderborg Hospital (Other Government)
Collaborators: The Danish Midwifery Organization (Unknown); Aase and Ejnar Danielsens Foundation (Other); The Augustinus Foundation, Denmark. (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11295
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-09

CONDITIONS: Birth Injuries; Lacerations; Pain
Keywords: Perineal; repair; episiotomies; midwives; pain relief; Episiotomy
MeSH Terms: conditions — Birth Injuries; Lacerations; Pain | interventions — Acupuncture Therapy; Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Procedure: acupuncture in 6 specific points
Drug: lidocaine 10mg/ml

SUMMARY:
Midwives and obstetricians are currently using acupuncture for several health problems during pregnancy and childbirth. The investigators wish to determine whether acupuncture can be used as pain relief during the repair of lacerations in the female pelvic floor following childbirth.

Three acupuncture points in the ear have been reported highly effective for perineal pain relief. A scientific trial will compare acupuncture with traditional local anaesthetics when midwives conduct perineal repair just after delivery in the hospitals of Southern Denmark.

DETAILED DESCRIPTION:
A randomised trial has been initiated. 226 healthy primipara are invited to participate if they deliver a child after gestation week 36 and sustain a perineal laceration or an episiotomy during childbirth.

The randomisation is done using a computer-controlled voice response system and the compared treatments are:

A: Acupuncture in Shen Men, GV20, BL36 and 2 needles in the upper ear.

B: Local anaesthetics (lidocaine 10 ml/mg) directly in the wound area.

Primary outcomes are:

1. Need for additional pain relief during the perineal repair.
2. Pain experienced during perineal repair reported 1 day after delivery.
3. Wound healing evaluated 1 and 14 days after delivery.
4. Patient satisfaction with the given pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Primipara
* Healthy mother and child
* Danish speaking
* Perineal laceration or episiotomy that can be sutured by a midwife.

Exclusion Criteria:

* Large perineal lacerations
* Heavy bleeding after childbirth
* No need for pain relief

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 207 (Actual)
Dates: Start 2006-05; Primary Completion 2007-07 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Need for additional pain relief during the perineal repair
Pain experienced during perineal repair reported 1 day after delivery
Wound healing evaluated 1 and 14 days after delivery

SECONDARY OUTCOMES:
Patient satisfaction with the given pain relief

CONTACTS AND LOCATIONS:
Overall Officials: Sara Kindberg, PhD Student, Principal Investigator — Aarhus University, Perinatal Epidemiological Unit
Locations (1):
- Obstetric Departments in the Hospitals of Southern Denmark, Sønderborg, Region Syddanmark, Denmark